CLINICAL TRIAL: NCT02395614
Title: Post-Mastectomy Surgical Pocket Irrigation With Triple Antibiotic Solution vs Chlorhexidine Gluconate: A Randomized Controlled Trial Assessing Surgical Site Infections in Immediate Tissue Expander Breast Reconstruction
Brief Title: Surgical Site Infection With 0.05% Chlorhexidine (CHG) Compared to Triple Antibiotic Irrigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Kent Higdon, MD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 140231
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
Keywords: tissue expander; breast reconstruction
MeSH Terms: conditions — Breast Neoplasms | interventions — Gentamicins; Cefazolin; Bacitracin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine irrigation (Experimental): 0.05% chlorhexidine solution (IrriSept®) commercially prepared in 450 ml bottles for irrigation. Each patient will receive triple antibiotic solution on one breast and the CHG on the other breast.
  Interventions: Drug: Chlorhexidine irrigation
- triple antibiotic irrigation (Active Comparator): triple antibiotic solution will contain 1 g of cefazolin, 50,000 U of bacitracin, and 80 mg of gentamicin in 500 mL of normal saline (NS). If the patient is allergic to either component - the allergen will not be used in the solution - for irrigation. Each patient will receive triple antibiotic solution on one breast and the CHG on the other breast.
  Interventions: Drug: triple antibiotic irrigation

INTERVENTIONS:
Drug: Chlorhexidine irrigation — - 0.05% chlorhexidine solution (IrriSept®) commercially prepared in 450 ml bottles will be used to irrigate one breast pocket. Each patient will receive triple antibiotic solution on one breast and the CHG on the other breast.
  Other Names: CHG
  Arms: Chlorhexidine irrigation
Drug: triple antibiotic irrigation — -triple antibiotic solution will contain 1 g of cefazolin, 50,000 U of bacitracin, and. Each patient will receive triple antibiotic solution on one breast and the CHG on the other breast.
  80 mg of gentamicin in 500 mL of NS. If the patient is allergic to either component - the allergen will not be used in the solution - to irrigate one breast pocket
  Other Names: gentamicin, cefazolin and bacitracin
  Arms: triple antibiotic irrigation

SUMMARY:
The investigators intend to perform a prospective randomized study and compare the incidence of surgical wound infection between mastectomy wounds irrigated with triple antibiotic solution (one side) and 0.05% CHG (opposite side) in patients undergoing bilateral breast reconstruction. Each patient will receive triple antibiotic solution on one breast and the CHG on the other breast.

DETAILED DESCRIPTION:
Breast reconstruction with tissue expander (TE) remains the gold standard of breast restoration after mastectomy. During the first stage of reconstruction, a TE is placed under chest muscles and slowly inflated postoperatively over the period of several weeks. After desired volume of TE is achieved it is exchanged for permanent breast prosthesis during another surgery (second stage of reconstruction). Postoperative wound infection after placement of TE can lead to devastating consequences both for patients and a surgeon. Frequently, surgical site infection requires additional surgeries and resulting in the removal of TE and long term IV antibiotic therapy. Therefore, during breast reconstruction procedures all possible measures are implemented to reduce postoperative infection rate. Several studies demonstrated that intra-operative irrigation of surgical wounds with antibiotic containing solution before insertion of breast TE decreases postoperative infection rate. This approach is currently adopted as a standard of care within plastic surgery clinical community.

The investigators intend to perform a prospective randomized study and compare the incidence of surgical wound infection between mastectomy wounds irrigated with triple antibiotic solution (one side) and 0.05% CHG (opposite side) in patients undergoing bilateral breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* females between 18 - 81 years of age
* and are undergoing bilateral mastectomy
* and are candidates for immediate breast reconstruction with tissue expanders.

Exclusion Criteria:

* females younger than 18 and older than 81 years of age;
* undergoing unilateral mastectomy and reconstruction;
* bilateral reconstruction using other techniques,
* patients allergic to one or more components of the antibiotic solution;
* allergy to CHG

Ages: 18 Years to 81 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-12; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Higdon, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Undergoing Bilateral Mastectomy: This group includes participants undergoing bilateral mastectomy with immediate breast reconstruction and tissue expander.
  Each participant will receive an irrigation of chlorhexidine solution 0.05% (IrriSept, 0.05% CHG in sterile water) on one breast and an irrigation of triple antibiotic solution (composed of cefazolin, gentamicin, and bacitracin) on the other breast.
Period: Overall Study
Arm/Group | Participants Undergoing Bilateral Mastectomy
Started | 88
Chlorhexidine Irrigation | 88
Triple Antibiotic Irrigation | 88
Completed | 88
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: 88 participants were included. In each participant, 1 mastectomy pocket was randomized to TAS and the other to CHG.
  CHG consisted of commercially prepared 0.05% CHG solution (IrriSept, 0.05% CHG in sterile water, IrrimaxCorporation, Lawrenceville, GA).
  TAS contained 1 g of cefazolin, 50,000 U of bacitracin, and 80 mg of gentamicin in 500 mL of normal saline.
Arm/Group | All Participants
Number analyzed (Participants) | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 88
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Females | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 81
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 88
BMI [Mean (Inter-Quartile Range); unit: kg/m^2] | 28.2 [23.5 to 32.4]
Tobacco use [Count of Participants; unit: Participants] | 4
Comorbidities [Count of Participants; unit: Participants]
  Diabetes | 5
  Hypertension | 15
  DVT | 2
  Bleeding disorders | 2
  No comorbidities | 64
Indication for mastectomy [Count of Participants; unit: Participants]
  Unilateral cancer | 71
  Bilateral cancer | 5
  Bilateral risk reducing | 12
Cancer treatment [Count of Participants; unit: Participants]
  Neoadjuvant therapy | 2
  Adjuvant radiation | 10
  Chemotherapy | 35
  None | 41
Alcohol use [Count of Participants; unit: Participants] | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Site Infection
Description: At all postoperative visits with the reconstructive surgeon, patients were thoroughly examined for presence of SSI (cellulitis, purulent drainage). SSI was defined as any instance where antibiotics were restarted or where erythema, cellulitis, warmth, purulent drainage, or fever occurred. SSI was further classified in 3 categories: minor when requiring oral antibiotics, major when requiring inpatient intravenous antibiotics or operative washout, and finally, explantation.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Participants Undergoing Bilateral Mastectomy
Number analyzed (Participants) | 88
participants
  Chlorhexidine irrigation | 7
  Triple antibiotic irrigation | 4

2. Secondary Outcome: Number of Participants With Flap Necrosis, Hematoma, and Seroma
Description: At all postoperative visits with the reconstructive surgeon, patients were thoroughly examined for presence of necrosis, seroma, or hematoma.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Participants Undergoing Bilateral Mastectomy
Number analyzed (Participants) | 88
participants
  Chlorhexidine irrigation | 21
  Triple antibiotic irrigation | 23

ADVERSE EVENTS:
Time Frame: 20 months
Groups:
- Chlorhexidine Irrigation: Each patient received triple antibiotic solution on one breast and the CHG on the other breast.
  CHG consisted of commercially prepared 0.05% CHG solution (IrriSept, 0.05% CHG in sterile water, Irrimax Corporation, Lawrenceville, GA.
- Triple Antibiotic Irrigation: Each patient received triple antibiotic solution on one breast and the CHG on the other breast.
  Triple antibiotic solution contains 1 g of cefazolin, 50,000 U of bacitracin, and 80 mg of gentamicin in 500 mL of normal saline (NS). If the patient is allergic to either component - the allergen will not be used in the solution - for irrigation.
Arm/Group | Chlorhexidine Irrigation | Triple Antibiotic Irrigation
All-Cause Mortality (participants affected / at risk) | 2/88 | 2/88
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/88
Other Adverse Events (participants affected / at risk) | 33/88 | 29/88
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chlorhexidine Irrigation (N=88) | Triple Antibiotic Irrigation (N=88)
Surgical site infections (Infections and infestations) | 7 | 4
Necrosis/Hematoma/Seroma (Blood and lymphatic system disorders) | 21 | 23
Explantation secondary to infection (Infections and infestations) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-04-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT02395614/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT02395614/ICF_001.pdf